CLINICAL TRIAL: NCT00680550
Title: Indications for Diagnosis, Arrhythmia and Monitoring of Reveal XT.
Brief Title: INSIGHT (R)XT. Indications for Diagnosis, Arrhythmia and Monitoring of Reveal XT
Status: Completed | Type: Observational
Sponsor: Medtronic BRC (Industry)
Responsible Party: Sponsor
Other Study IDs: CMD 466
Record Dates: First submitted 2008-05-15; First posted 2008-05-20 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Atrial Fibrillation; Cardiac Arrhythmias
Keywords: Atrial Fibrillation; Risk of cardiac Arrhythmias; Loop recorder
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To describe the clinical indications for Reveal XT in diagnosis and continuous monitoring of arrhythmia and to explore the clinical applications and outcome of arrhythmia monitoring on patient care.

DETAILED DESCRIPTION:
Improving the diagnosis and management of cardiac rhythm disturbances remains a major challenge for physicians. Limitations of current cardiac arrhythmia monitoring using ECG, holters or event recorders are that these methods are non-continuous and/or automatic arrhythmia detection is often impossible. The Medtronic Reveal XT Insertable Cardiac Monitor is a programmable device which continuously monitors the patient's subcutaneous ECG and provides information regarding arrhythmia episodes, long term trending of AF burden, patient's activity and heart rate variability. The Reveal XT records cardiac information in response to patient activation and automatically detected arrhythmias thereby offering advantages over conventional tools for long-term arrhythmia monitoring with regard to compliance and recording time.

The clinical applications for Reveal XT are varied. Diagnostic, arrhythmia monitoring and arrhythmia management functions can be discriminated.

This study is a prospective, observational, multicenter international post-market study. The results of this study will describe the different patient groups for which the Reveal XT is being used for the diagnosis and monitoring of various cardiac arrhythmias. This study will also collect data regarding the clinical consequences of using the Reveal XT and the influence of Reveal XT data on clinical care pathways. The physician as well as the patient's satisfaction with the device will be evaluated. The study will be conducted in 60-100 centers primarily in Europe. It is expected that 800-1000 patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Patient implanted or scheduled for an implant with a Reveal XT Insertable Cardiac Monitor System for arrhythmia diagnosis or monitoring
* Patient must be willing to sign a Patient Data Release Form (or Informed Consent where applicable)

Exclusion Criteria:

* Enrollment outside a 30-day window from the planned/performed Reveal XT implant procedure (from 15 days pre-implant until 15 days post implant)
* Patient is implanted with a pacemaker, ICD, CRT-device or an implantable hemodynamic monitoring system
* Unwillingness or inability to cooperate or give written informed consent or, if the patient is a minor and the legal guardian refuses to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients currently implanted with, or who will be implanted with a Reveal XT Insertable Cardiac Monitor for arrhythmia diagnosis or monitoring.
Sampling Method: Probability Sample
Enrollment: 1003 (Actual)
Dates: Start 2008-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
descriptive: clinical indications for Reveal XT | 2008-2012
  To describe the patient population implanted with a Reveal XT for arrhythmia diagnosis and monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Guido Rieger, MD, Study Chair — Medtronic Bakken Research Center BV
Locations (56):
- Austria (3):
  - Krankenhaus der Elisabethinen, Linz
  - Universitätsklinik für Innere Medizin, Vienna
  - Klinkum Wels-Grieskirchen GmbH, Wels
- Republican Scientific Practical Center, Minsk, Belarus
- Czechia (3):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - Kardiologicka ambulance, Ostrava
- Tampere University Hospital, Tampere, Finland
- Germany (23):
  - Zentralklinik Bad Berka, Bad Berka
  - St.-Marien-Hospital, Bonn-Venusberg
  - Kardiologische Praxis, Burg
  - Klinikum Coburg, Coburg
  - Kardiologische Praxis, Dessau
  - Herzzentrum Dresden, Dresden
  - Kardiocentrum, Frankfurt
  - Universitatsklinikum, Freiburg im Breisgau
  - St. Johannes Hospital, Hagen
  - Universitares Herzzentrum, Hamburg
  - Medizinische Hochshule, Hanover
  - Asklepios Klinik, Harburg
  - Uniklinik Homburg - Klinik fur Innere Medizin III, Homburg
  - Herzzentrum, University of Leipzig, Leipzig
  - Klinik Augustinum, München
  - Klinikum der Universität München-Großhadern (LMU), München
  - Universitätsklinikum Münster, Münster
  - Klinikum Nürnberg Süd, Nuremberg
  - St. Martinus Hospital, Olpe
  - DRK-Krankenhaus Mölln-Ratzeburg, Ratzeburg
  - Krankenhaus Barmherzige Brueder, Regensburg
  - Krankenhaus Reinbek, St.-Adolf-Stift, Reinbek
  - Universitaetsklinikum Tuebingen, Tübingen
- Azienda Ospedaliera Universitaria Careggi, Florence, Italy
- Netherlands (8):
  - Gelre Apeldoorn, Apeldoorn
  - Ziekenhuis De Tjongerschans, Heerenveen
  - Bethesda Ziekenhuis, Hoogeveen
  - Westfries Gasthuis, Hoorn
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Vlietland Ziekenhuis, Schiedam
  - Maasland Ziekenhuis, Sittard
  - Diakonessenhuis Utrecht, Utrecht
- Centro Hospitalar do Porto - Hospital de Santo Antonio, Porto, Portugal
- Russia (4):
  - Scientific Research Center of Cardio Vascular Surgery by A.N. Bakulev, Moscow
  - State Research Institute of Circulation Pathology, Novosibirsk
  - Almazov Federeal Heart, Blood and Endocrinology Centre, Saint Petersburg
  - Tyumen Cardiology Centre, Tyumen
- Arytmologicke oddelenie VUSCH, Košice, Slovakia
- University Medical Center Ljubljana, Ljubljana, Slovenia
- Complejo Hospitalario Universitario de Vigo, Vigo, Spain
- University Hospital Örebro, Örebro, Sweden
- Switzerland (5):
  - Hopital Cantonal de Fribourg, Fribourg
  - Hopital Cantonal Universitaires de Geneve, Geneva
  - Hopital de Pourtales de Neuchatel, Neuchâtel
  - Hopital de Sion CHCVS, Sion
  - UniversitatsSpital, Zurich
- Sheikh Khalifa Medical Center, Abu Dhabi, United Arab Emirates
- Liverpool Heart and Chest Hospital, Liverpool, United Kingdom